CLINICAL TRIAL: NCT06293157
Title: Carbon Fiber Transpedicular Screws in Treatment of Spinal Metastatic Disease and Stereotactic Radiotherapy - a Prospective, Randomized Trial
Brief Title: Carbon Fiber Transpedicular Screws in Treatment of Spinal Metastatic Disease
Acronym: CarboMetaspine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copernicus Memorial Hospital (Other)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Principal Investigator, Kamil Krystkiewicz, Principal Investigator, Copernicus Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/ABM/01/00013
Record Dates: First submitted 2024-02-17; First posted 2024-03-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Spinal Cord Compression; Metastasis Spine
Keywords: metastatic spinal disease; stereotactic body radiotherapy; spinal cord compression; carbon fiber reinforced implants
MeSH Terms: conditions — Spinal Cord Compression; Spinal Diseases | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transpedicular spinal stabilization using carbon system + SBRT (Experimental): Transpedicular spinal stabilization using a radiolucent composite system made of carbon fibers and PEEK followed by stereotactic radiotherapy of the spine at a dose of 5x5 Gy (25 Gy in the total dose)
  Interventions: Procedure: Transpedicular spinal stabilization - carbon fibers-based implants; Radiation: Stereotactic body radiotherapy
- Transpedicular spinal stabilization using titanium system + SBRT (Active Comparator): Transpedicular spinal stabilization using a titanium system followed by stereotactic radiotherapy of the spine at a dose of 5x5 Gy (25 Gy in the total dose)
  Interventions: Procedure: Transpedicular spinal stabilization - titanium implants; Radiation: Stereotactic body radiotherapy
- SBRT + Transpedicular spinal stabilization using titanium system (Sham Comparator): Transpedicular spinal stabilization using a titanium system preceded with stereotactic spine radiotherapy at a dose of 5x5 Gy (25 Gy in the total dose) as the first stage of treatment
  Interventions: Procedure: Transpedicular spinal stabilization - titanium implants; Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Procedure: Transpedicular spinal stabilization - carbon fibers-based implants — Transpedicular stabilization with carbon fiber and PEEK-based implants in one of the two possible variants - first involves a large skin incision and separation of the back extensor muscles; second is associated with minimally invasive, which is percutaneous procedure that allows the stabilization with implants without the need to detach the muscles, using only a small skin incision.
  Arms: Transpedicular spinal stabilization using carbon system + SBRT
Procedure: Transpedicular spinal stabilization - titanium implants — Transpedicular stabilization with titanium implants in one of the two possible variants - first involves a large skin incision and separation of the back extensor muscles; second is associated with minimally invasive, which is percutaneous procedure that allows the stabilization with implants without the need to detach the muscles, using only a small skin incision.
  Arms: SBRT + Transpedicular spinal stabilization using titanium system; Transpedicular spinal stabilization using titanium system + SBRT
Radiation: Stereotactic body radiotherapy — Spinal tumors will be treated with stereotactic body radiotherapy at a dose of 5x5 Gy (25 Gy in a total dose); either prior to or post-surgical treatment, accordingly the allocation to one of the study arms.
  Other Names: SBRT

SUMMARY:
Background: Spinal metastatic disease constitute a serious clinical problem in oncology. Bones are the third most common organ where metastases are located, and the spine is the place where they are most often located. Due to the complexity of the clinical problem, metastatic spine disease remains of interest to many medical specialties: neurosurgery, orthopedics, clinical oncology, radiotherapy and rehabilitation. With the development of modern diagnostic methods and wider access to them, the demand for neurosurgical treatment in this group of patients is growing. Surgical treatment is undertaken in cases of spinal cord compression, instability, spinal deformation or pain that is resistant to radiotherapy. The standard treatment in most cases is posterior instrumentation of the spine using titanium pedicle screws. Unfortunately, these systems cause numerous artifacts in diagnostic imaging, both in CT and MRI. These distortions make it difficult to plan radiotherapy and determine the optimal dose that would avoid healthy tissues. Moreover, artifacts could make difficult postoperative follow-ups aimed at assessing local recurrence. The solution to these problems is the use of radiolucent implants. There are systems based on carbon fibers embedded in PEEK which do not cause typical artifacts for titanium implants.

Study plan: The open, three-arm, prospective randomized study is planned to involve 226 patients with metastatic disease of the spine, with a known or undiagnosed primary site. Patients will be qualified for 2 types of interventions. The first one includes treatment with stereotactic radiotherapy (SBRT) in the first stage of treatment and early instrumentation of the spine with titanium implants. The second type of intervention includes patients qualified for surgical treatment using spine stabilization and postoperative SBRT. Patients within this arm will be randomized into two groups differing in the type of material the instrumentation is made of: carbon-PEEK or titanium. The study group will be patients stabilized with carbon implants, and the control group will be those who will have titanium implants.

Study population: The study includes adult patients with metastatic spine disease, with a known or unknown primary tumor, qualified for SBRT and surgical treatment.

Assumed effects: It is assumed that the treatment proposed in the project would extend progression free survival by several months or achieve local control in an additional 5% of patients. Moreover, by improving the quality of imaging, earlier diagnosis of local recurrences and implementation of appropriate locoregional treatment would be possible.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic spinal disease,
* ECOG quality of life of 0-2,
* Eligibility for SBRT treatment,
* Expected survival time >3 months,
* Signed informed consent to participate in the study,
* Sufficient organ capacity allowing to survive the perioperative period.

Exclusion Criteria:

* Primary tumor of the spine,
* Age <18 years old,
* Expected survival time <3 months,
* Eligibility for palliative radiotherapy,
* No informed consent to participate in the study,
* Pregnancy or breastfeeding,
* The advancement of the disease preventing the technical use of implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
The assessment of time to local recurrence after treatment with SBRT. | 5 years
The assessment of frequency of local recurrence after treatment with SBRT. | 5 years

SECONDARY OUTCOMES:
DICE convergence factor evaluation between groups of patients. | 1 day
  The use of convergence factor assessment will allow for comparison of similarity in planned SBRT between all groups. This will allow an indirect assessment of difficulties in planning treatment by a radiotherapist using objective tools.
The subjective difficulty of planning radiotherapy treatment. | 1 day
  Using a numerical scale from 0-10, the radiotherapist will assess the difficulty of planning, tumor coverage, and delineation of the spinal cord depending on the group assessed in the study.
The frequency of radiation complications assessed according to the National Cancer Institute Common Toxicity Criteria (NCI CTC). | 5 years
  Titanium instrumentation generates significant artifacts in radiological imaging used for radiotherapy planning. The use of opaque, radiolucent material allows for radiotherapy planning to cover a smaller area. This may reduce the incidence of radiation-related complications in nearby organs (OAR - organ at risk). These complications will be assessed by the radiation therapist according to the standardized NCI CTC scale. Potentially smaller quantity of organ complications could be an advantage supporting the use of carbon implants.
Failure rate of stabilizing systems. | 5 years
  Titanium and carbon fiber show similar biocompatibility. The biomechanical properties of these materials are also similar. In vitro studies have shown a similar effect failure rate of carbon pedicle screws compared to standard titanium ones. However, carbon rods have greater flexibility and structure connected using these may show more frequent loosening in vivo, especially in cases with impaired sagittal balance. This was not an issue analyzed in the literature. The frequency of instrument failure is of great importance for clinical practice because most such cases require operative revision.
Pain assessment on the VAS scale between groups. | 5 years
  One of the goals of surgical treatment is to treat mechanical pain caused by segmental instability. SBRT is a good method of treating biological pain. There are no comparisons of analgesic effects between transpedicular systems. Greater pain reduction allows for more effective and longer ability to walk, lower consumption of painkillers, and lower incidence of complications related to immobilization (thrombosis, bedsores, respiratory infections), which also has pharmacoeconomic implications.
Frequency of postoperative infections. | 5 years
  Postoperative wound infections are an inherent complication of surgical procedures. The longer the procedure, the more often inflammatory complications are observed, especially in oncological population, which has a higher average age of treated patients, a greater number of burdens, frequent immunosuppression due to systemic treatment, and malnutrition in the form of decreased biochemical parameters (total protein and albumin). Titanium has good properties in this aspect. Bacterial biofilms, is rarely formed on it, which means that patients can be treated more often without the need to remove the implants. It is unclear how carbon fiber system will perform in these cases. There are not made of metal, but of carbon fiber embedded in polymer. Assessment of the frequency of inflammatory complications and their course will provide the answer to whether This instrumentation allows for a similar management strategy in clinical settings.
Differences in dosimetric parameter Dmin PTV/CTV. | 1 day
Differences in dosimetric parameter D95. | 1 day
Differences in dosimetric parameter D98. | 1 day
Differences in dosimetric parameter D100. | 1 day
Differences in dosimetric parameter conformity index (CI) / homogeneity index (HI)). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Krystkiewicz, PhD, Principal Investigator — Department of Neurosurgery and Neurooncology, Copernicus Memoriał Hospital in Łódź
Locations (5):
- Poland (5):
  - Department of Neurosurgery, Functional Neurosurgery and Stereotaxy, Dr. Jan Biziel University Hospital No. 2 in Bydgoszcz, Bydgoszcz
  - Professor Franciszek Łukaszczyk Oncology Center in Bydgoszcz - National Research Institute, Bydgoszcz
  - Department of Teleradiotherapy, Lower Silesian Center of Oncology, Pulmonology and Hematology, Wroclaw
  - University Center of Neurology and Neurosurgery, Jan Mikulicz-Radecki University Clinical Hospital in Wrocław, Wroclaw
  - Copernicus Memorial Hospital in Łódź, Poland, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cofano F, Di Perna G, Monticelli M, Marengo N, Ajello M, Mammi M, Vercelli G, Petrone S, Tartara F, Zenga F, Lanotte M, Garbossa D. Carbon fiber reinforced vs titanium implants for fixation in spinal metastases: A comparative clinical study about safety and effectiveness of the new "carbon-strategy". J Clin Neurosci. 2020 May;75:106-111. doi: 10.1016/j.jocn.2020.03.013. Epub 2020 Mar 12. PMID 32173153
- [Background] Boriani S, Tedesco G, Ming L, Ghermandi R, Amichetti M, Fossati P, Krengli M, Mavilla L, Gasbarrini A. Carbon-fiber-reinforced PEEK fixation system in the treatment of spine tumors: a preliminary report. Eur Spine J. 2018 Apr;27(4):874-881. doi: 10.1007/s00586-017-5258-5. Epub 2017 Aug 16. PMID 28815357
- [Background] Nevelsky A, Borzov E, Daniel S, Bar-Deroma R. Perturbation effects of the carbon fiber-PEEK screws on radiotherapy dose distribution. J Appl Clin Med Phys. 2017 Mar;18(2):62-68. doi: 10.1002/acm2.12046. Epub 2017 Feb 7. PMID 28300369
- [Background] Ringel F, Ryang YM, Kirschke JS, Muller BS, Wilkens JJ, Brodard J, Combs SE, Meyer B. Radiolucent Carbon Fiber-Reinforced Pedicle Screws for Treatment of Spinal Tumors: Advantages for Radiation Planning and Follow-Up Imaging. World Neurosurg. 2017 Sep;105:294-301. doi: 10.1016/j.wneu.2017.04.091. Epub 2017 May 3. PMID 28478252
- [Background] Neal MT, Richards AE, Curley KL, Patel NP, Ashman JB, Vora SA, Kalani MA. Carbon fiber-reinforced PEEK instrumentation in the spinal oncology population: a retrospective series demonstrating technique, feasibility, and clinical outcomes. Neurosurg Focus. 2021 May;50(5):E13. doi: 10.3171/2021.2.FOCUS20995. PMID 33932921
- [Background] Lindtner RA, Schmid R, Nydegger T, Konschake M, Schmoelz W. Pedicle screw anchorage of carbon fiber-reinforced PEEK screws under cyclic loading. Eur Spine J. 2018 Aug;27(8):1775-1784. doi: 10.1007/s00586-018-5538-8. Epub 2018 Mar 1. PMID 29497852

DOCUMENTS (1):
  • Informed Consent Form (2025-05-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT06293157/ICF_002.pdf